CLINICAL TRIAL: NCT01036139
Title: A Randomized, Multicenter 12-Week Double-blind Placebo-controlled Study to Assess the Efficacy and Safety of BF2.649 in Excessive Daytime Sleepiness in Parkinson's Disease Followed by a 38-Week Open-label Extension Phase
Brief Title: Efficacy and Safety of BF2.649 in Excessive Daytime Sleepiness (EDS) in Parkinson's Disease
Acronym: HARPS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06-10 / BF 2.649; Eudract number (Other: 2009-013885-14)
Record Dates: First submitted 2009-12-11; First posted 2009-12-21 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Parkinson's Disease
Keywords: EDS in Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF2.649 (pitolisant) (Experimental): BF2.649 (5mg, 10 mg, 20 mg) in capsules
  Interventions: Drug: BF2.649 (pitolisant)
- Placebo (Placebo Comparator): Placebo of BF2.649 (5mg, 10mg, 20mg) in capsules
  Interventions: Drug: BF2.649 (pitolisant)

INTERVENTIONS:
Drug: BF2.649 (pitolisant) — 1 capsule of BF2.649 (5mg, 10mg , 20 mg) O.D
  Other Names: Pitolisant

SUMMARY:
To compare the efficacy of BF2.649 over placebo (12 week Double-Blind Phase) and assess the long term safety and the efficacy maintenance(9 months Open-Label Extension Phase) of BF2.649 in the improvement of excessive daytime sleepiness in patients diagnosed with Parkinson's Disease.

DETAILED DESCRIPTION:
As measured by the change from baseline in the Epworth Scale Scores (ESS) at Week 12 and at Week 51, in patients diagnosed with EDS in Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented history of Parkinson's disease according to UPDRS,fluctuating and non-fluctuating patients, Hoehn and Yahr score <5;
* stabilized on optimal antiparkinsonian treatments unmodified for 4 weeks prior to study entry;
* presenting an Excessive Daytime Sleepiness as indicated by an ESS>or=12

Exclusion Criteria:

* Patients with a known diagnosis of other degenerative parkinsonian syndromes (e.g. Progressive supra-nuclear palsy, multisystemic atrophy, corticobasal degenerescence, diffuse Lewy's Body dementia)
* Patients who have shift work, chronic or occasional sleep deprivation, circadian rhythm disorders
* Patients with a severe depression indicated by (BDI>= 16)or at suicidal risk (BDI item G>0) or depression treated for less than 8 weeks
* Patients with a cognitive impairment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
ESS change (Epworth Sleepiness Scale) | at week 12 / 52 versus baseline

SECONDARY OUTCOMES:
Safety | 12-week and 52-week
  Any AE observed and reported during the study

CONTACTS AND LOCATIONS:
Overall Officials: Kati Gutierrez, PharmD, Study Director — Bioprojet
Locations (1):
- Pr Arnulf, Paris, France